CLINICAL TRIAL: NCT06580964
Title: Glycemic Control and Frailty Risk in Older People at Risk for Type 2 Diabetes: Impact of Local Heat Therapy
Brief Title: Heat and Exercise in Aging as Therapy (HEAT)
Acronym: HEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01AG084597 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Prediabetic State
Keywords: Exercise; Heat; Aging; Prediabetes; Skeletal Muscle
MeSH Terms: conditions — Prediabetic State; Motor Activity | interventions — Diathermy; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Local Heat Therapy (Experimental): Phase 1: Heat pads will be applied to both legs and set to a pre-determined, optimized temperature to raise the intramuscular temperature to 3-4°C above resting. Each heating session will last for 90 min/d, 6d/wk (5 at-home and 1 in-lab) for 12 wks.
  Phase 2: High-intensity interval training will be performed 3 d/wk for 12 wks. Each exercise session will consist of 4 cycling exercise intervals (4 min each) with 3 min active rest between intervals. Interval intensity will progressively increase from 70-75% to 90-95% of VO2peak by the end of week 3.
  Interventions: Behavioral: Heat therapy; Behavioral: High-intensity interval training
- Thermoneutral Therapy (Sham Comparator): Phase 1: Heat pads will be applied to both legs and set to a pre-determined temperature to keep the intramuscular temperature in a thermoneutral state (~35-37°C). Each heating session will last for 90 min, 7d/wk (6 at-home and 1 in-lab) for 12 weeks.
  Phase 2: High-intensity interval training will be performed 3 d/wk for 12 wks. Each exercise session will consist of 4 cycling exercise intervals (4 min each) with 3 min active rest between intervals. Interval intensity will progressively increase from 70-75% to 90-95% of VO2peak by the end of week 3.
  Interventions: Behavioral: Heat therapy; Behavioral: High-intensity interval training
- High-Intensity Interval Training (Active Comparator): Phase 1: High-intensity interval training will be performed 3 d/wk for 12 wks. Each exercise session will consist of 4 cycling exercise intervals (4 min each) with 3 min active rest between intervals. Interval intensity will progressively increase from 70-75% to 90-95% of VO2peak by the end of week 3.
  Phase 2: N/A.
  Interventions: Behavioral: High-intensity interval training

INTERVENTIONS:
Behavioral: Heat therapy — Heat pads will be set to a pre-determined, optimized temperature and applied to both legs for 90 min, 6d/wk (5 at-home and 1 in-lab).
  Arms: Local Heat Therapy; Thermoneutral Therapy
Behavioral: High-intensity interval training — High-intensity interval training will be performed 3 days per week for 12 weeks.

SUMMARY:
The main goal of this two-phase clinical trial is to learn whether local heat therapy, using heat pads applied to the legs, can enhance skeletal muscle health, physical function, and blood sugar control in a manner comparable to exercise, specifically High-Intensity Interval Training (HIIT), in older individuals with prediabetes. The study aims to answer the following questions:

1. Does local heat therapy improve muscle architecture (e.g., muscle cross-sectional area, capillary density, mitochondrial content), glucose tolerance, and frailty indicators similarly to HIIT in older individuals with prediabetes?
2. Does local heat therapy as a pre-conditioning method enhance the skeletal muscle response to HIIT in older individuals with prediabetes?

DETAILED DESCRIPTION:
To achieve the study objectives, researchers will first compare the outcomes of local heat therapy to: 1) HIIT and 2) heat pads set to maintain normal skeletal muscle temperature (control group). Then, researchers will compare the outcomes of the local heat therapy and control groups after a subsequent HIIT intervention. This will enable the researchers to assess the effectiveness of local heat therapy (compared to HIIT and preceding HIIT) to improve skeletal muscle health, physical function, blood sugar control.

Study Procedures:

All participants will visit the laboratory over three days at the start of the study for baseline assessments and sample collection.

Participants in the Control (CON) and Local Heat Therapy (LHT) groups will:

Phase 1:

* Use heat pads on both thighs at a pre-determined temperature for 90 minutes daily, 6 days a week (5 days at home and 1 day in the laboratory; 12 laboratory visits) for the first 12 weeks.
* Maintain a log of each heat pad session.
* Visit the laboratory over three days at the end of Phase 1 for follow-up assessments and sample collection.

Phase 2:

* Visit the laboratory three days per week for 12 weeks (a total of 36 visits) for exercise training.
* Visit the laboratory over three days at the end of Phase 2 for final assessments and sample collection.

Participants in the HIIT Group will:

Phase 1:

* Visit the laboratory three days per week for 12 weeks (a total of 36 visits) for exercise training.
* Visit the laboratory over three days at the end of Phase 1 for final assessments and sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Women who are postmenopausal, defined as no menstrual period for at least 12 consecutive months.
* Sedentary (structured exercise <30 minutes, 3x/week)
* Body weight is at least 110 lbs
* Meet criteria for prediabetes (fasting blood glucose 100-125 mg/dl, hemoglobin A1c 5.7-6.4%)
* Consume <8 (women) or <15 (men) alcohol-containing beverages per week
* Do not use nicotine or cannabis
* Not taking any medications that could interfere with responses to the interventions (e.g., corticosteroids, opiates, benzodiazepines, tricyclic antidepressants, beta blockers, sulfonylureas, insulin, metformin, anticoagulants, barbiturates, insulin sensitizers, fibrates, immunosuppressants). If you don't know, that's okay. We'll ask what medications you are on and check whether they fall into one of these categories.

Exclusion Criteria:

* History of peripheral neuropathies
* Currently taking prescription blood thinners
* Medical complications that could would contraindicate participation in the high intensity interval training (HIIT) intervention including: orthopedic complications that would limit your ability to perform cycling exercise, significant cardiovascular impairments (e.g., history of arrhythmias, severe uncontrolled hypertension, etc.), diagnosed metabolic disease (e.g., diabetes), renal disease, sickle cell anemia, or cancer in remission for <6 months.
* Known history of slow wound healing
* Lidocaine allergy
* Latex allergy
* Currently pregnant
* >1.5" subcutaneous fat over the thigh muscle
* Symptoms suggestive of cardiovascular, respiratory, metabolic, or renal diseases including discomfort, pressure, or pain in your chest, neck, jaw, arms, calves, or other areas potentially related to ischemia; shortness of breath at rest or with mild exertion; dizziness or fainting (syncope); difficulty breathing while lying flat (orthopnea) or sudden nighttime breathing difficulties (paroxysmal nocturnal dyspnea); palpitations or rapid heartbeat (tachycardia); pain or cramping in your legs during physical activity (intermittent claudication); a known heart murmur; swelling in your ankles (edema); unusual fatigue or shortness of breath during routine activities or at rest.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | Before intervention, after Phase 1 (at about 12 weeks), and after Phase 2 (at about 24 weeks, except HIIT group)
  Oral glucose tolerance test (OGTT)
Skeletal muscle architecture 1 | Before intervention, after Phase 1 (at about 12 weeks), and after Phase 2 (at about 24 weeks, except HIIT group)
  Immunohistochemical assessment of muscle fiber cross-sectional area and capillary density
Skeletal muscle architecture 2 | Before intervention, after Phase 1 (at about 12 weeks), and after Phase 2 (at about 24 weeks, except HIIT group)
  Assessment of skeletal muscle mitochondrial content
Frailty status | Before intervention, after Phase 1 (at about 12 weeks), and after Phase 2 (at about 24 weeks, except HIIT group)
  Fried's Phenotypic Frailty assessment
Exercise capacity | Before intervention, after Phase 1 (at about 12 weeks), and after Phase 2 (at about 24 weeks, except HIIT group)
  VO2peak testing

SECONDARY OUTCOMES:
Anthropometrics 1 | Weekly for about 14 (HIIT group) or about 27 (LHT and CON groups) weeks
  Body mass and height to calculate body mass index (BMI)
Anthropometrics 2 | Weekly for about 14 (HIIT group) or about 27 (LHT and CON groups) weeks
  Waist-to-hip ratio
Body composition | Before intervention, after Phase 1 (at about 12 weeks), and after Phase 2 (at about 24 weeks, except HIIT group)
  Lean versus fat mass assessed by dual-energy x-ray absorptiometry (DEXA)
Sleep quality | Weekly for about 14 (HIIT group) or about 27 (LHT and CON groups) weeks
  7-point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ying Luk, PhD; Danielle Levitt, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All raw data generated from this project will be stored on cloud-based servers at Texas Tech University. Cleaned data in an analysis-ready format will be stored in REDCap and periodically uploaded to repositories. Data of sufficient quality from human participants will be uploaded the Aging Research Biobank to allow others to validate replicate research findings.
  In alignment with the Data Submission Worksheet for the Aging Research Biobank, the following will be submitted to accompany deidentified data derived from human participants:
  * Full study protocol
  * Names and descriptions of data sets
  * Manual of operations
  * Annotated data collection forms
  * Data dictionary
  * Documentation of calculated variables
  * Summary of deidentification and crosslinking of study ID with new randomized ID
  * Any changes made to the protocol over time
  * Frozen datasets used for the primary publication, when applicable
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data associated with each publication will be made available when preprints are available and will continue to be available on the repositories and long as they are supported. Any data that are not yet available by the end of the award period will be made available at that time.
Access Criteria: Requests for data must be submitted through the Aging Research Biobank (see https://agingresearchbiobank.nia.nih.gov/how-to-make-a-request/).
URL: https://agingresearchbiobank.nia.nih.gov/